CLINICAL TRIAL: NCT02063789
Title: Prospective, Non-Randomized, Open-label, Single-arm, Multi-Center Phase III Clinical Trial to Evaluate the Efficacy and Safety of IV-Globulin SN Inj.10% in the Patients Diagnosed With Immune Thrombocytopenia (ITP).
Brief Title: An Open Phase 3 Study of IV-Globulin SN Inj.10% to Treat Immune Thrombocytopenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC5107A_P3
Record Dates: First submitted 2014-02-13; First posted 2014-02-14 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Immune Thrombocytopenia
Keywords: Immune Thrombocytopenia; Immune Thrombocytopenic Purpura; Idiopathic Thrombocytopenic Purpura; Human Immunoglobulin; ITP; IVIg; IgIV; IV-Globulin SN Inj.
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Human immunoglobulin intravenous (Experimental): Human immunoglobulin intravenous; GC5107A (IV-Globulin SN Inj. 10%); Day 1: GC5107A, 1g/kg, intravenous Day 2: GC5107A, 1g/kg, intravenous; Starting infusion rate: 0.01mg/kg/min (1mg/kg/min) for first 15 minutes, and then 2-fold increase every 30 minutes by maximum 0.08ml/kg/min (8mg/kg/min). Dosing modification is allowed due to tolerance.
  Interventions: Drug: Human immunoglobulin intravenous

INTERVENTIONS:
Drug: Human immunoglobulin intravenous — After GC5107A Intravenous injection, evaluate platelet increase
  Other Names: GC5107A (IV-Globulin SN Inj. 10%)

SUMMARY:
Human immunoglobulin (Ig) is the most commonly used blood product. It has been well-defined the efficacy in patients with immunodeficiencies, Kawasaki disease, asthma and other immune diseases. It is expected that Ig 10% will improve the usefulness and safety profile compared to Ig 5% because it is expected the reduced hospitalization/treatment duration and less adverse events related to volume overload.

DETAILED DESCRIPTION:
GC5107A (IV-Globulin SN Inj. 10%) is a polyvalent intravenous human immunoglobulin G preparation. It is prepared from plasma collected from more than 1000 healthy blood donors and it expresses the large spectrum of antibody specificity.

ELIGIBILITY:
Inclusion Criteria:

* Given written informed consent
* Male or female aged ≥ 19
* Primary immune thrombocytopenia (ITP)
* Platelet <20x10^9 /L
* Patients who have taken adrenal cortical hormones and/or other immunosuppressive medications should maintain their stable doses before and during this study

Exclusion Criteria:

* Patients who have participate in other interventional study within 30 days
* Inability in written/verbal communication
* Engaged with an elective surgery
* Pregnant or breast-feeding women
* Women of childbearing potential who do not agree with contraception during this study
* Patients who had experienced any hypersensitivity or shock with study drug or active ingredient
* Refractory to immunoglobulin therapy
* Secondary immune thrombocytopenia

  * HIV-associated ITP
  * Lupus-associated ITP
  * Lymphproliferative disease
  * Hepatitis virus carrier
  * Other disease- or infection-associated ITP
* Drug-Induced ITP
* Hereditary thrombopenia (e.g., MYH9 disorders)
* Hemolytic anemia (Positive direct Coomb's test)
* Clinically significant abnormalities of immunoglobulin
* Immunoglobulin A Deficiency
* Immune disorders or deficiency
* Alcohol or drug abuse within 6 months
* Patients who had taken any medications which may effect platelet function or count for at least 2 days prior study entry
* Patients who had administrated with IVIg or anti-D immunoglobulin agents within 1 month
* Patients who had undergone a splenectomy within 2 months
* Clinically significant underlying disease or medical history at investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
% of patients who achieved the platelet count ≥ 50 x 10^9/L increase | within 7 days after intervention

SECONDARY OUTCOMES:
Duration from the achievement of platelet count ≥ 50 x 10^9/L increase to the loss | 4 weeks after intervention
% patient with response | 4 weeks after intervention
  Response (R): platelet count ≥ 30 x 10^9/L and at least 2-fold increase of the baseline count, confirmed on at least 2 separate occasions at least 7 days apart, and absence of bleeding.
% patient with complete response | 4 weeks after intervention
  Complete response (CR): platelet count >100 x 10^9/L, confirmed on at least 2 separate occasions at least 7 days apart, and absence of bleeding.
Duration of response | 4 weeks after intervention
  measured from the achievement of R to loss of R
Duration of complete response | 4 weeks after intervention
  measured from the achievement of CR to loss of CR
% patient with no response | 4 weeks after intervention
  No response (NR): platelet count < 30 x 10^9/l or less than 2-fold increase of baseline platelet count, confirmed on at least 2 separate occasions approximately 1 day apart, or bleeding.
Descriptive statistics of platelet count at each visit | 4 weeks after intervention
Haemorrhage severity rate at each visit | 4 weeks after intervention
  Haemorrhage severity score (HSS) system
Quality of Life (EQ-5D) | 4 weeks after intevention
Patient reported bleeding events | 12 weeks after intervention
Usage of rescue mediations | 4 weeks after intervention
  Rescue medications: Acetaminophen, antihistamines.
Adverse events | 12 weeks after intervention
Drug compliance | 2 days of intervention
Viral safety | Base line, 4 weeks and 12 weeks after intervention
Time to the achievement of platelet count ≥50x10^9/L increase | within 7 days after intervention

OTHER OUTCOMES:
Pharmacokinetics of GC5107A | 12 weeks after intervention
  Day 1(pre-dosing, post dosing), 2 (pre-dosing, post dosing), 4, 8, 15, 29, and 85

CONTACTS AND LOCATIONS:
Overall Officials: Doyeun Oh, M.D., Ph.D., Principal Investigator — CHA Bundang Medical Center; Chang-Hee Lee, M.D, Study Director — Green Cross Corporation
Locations (14):
- South Korea (14):
  - Chungnam National University Hospital, Daejeon
  - Daegu Catholic University Medical Center, Deagu
  - Chonnam National University Hwasun Hospital, Hwasun
  - Gachon University Gil Medical Center, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Pusan National University Hospital, Pusan
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - CHA Budang Medical Center, Seoul
  - Ewha Womans University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Seoul
  - Soon Chung Hyang University Hospital, Seoul
  - VHS Medical Center, Seoul

REFERENCES:
- [Derived] Hong J, Bang SM, Mun YC, Yhim HY, Lee J, Lim HS, Oh D; Korean GC IVIg Investigators. Efficacy and Safety of a New 10% Intravenous Immunoglobulin Product in Patients with Primary Immune Thrombocytopenia (ITP). J Korean Med Sci. 2018 Apr 24;33(19):e142. doi: 10.3346/jkms.2018.33.e142. eCollection 2018 May 7. PMID 29736158